CLINICAL TRIAL: NCT00627315
Title: Prospective Study of Hormone Levels and Appetite After Bariatric Surgery
Brief Title: Prospective Study of Hormone Levels After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Judith Korner, Associate Professor of Medicine, Columbia University
Other Study IDs: AAAB0528; R01DK072011 (NIH)
Record Dates: First submitted 2008-02-28; First posted 2008-03-03 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Obesity
Keywords: Obesity; Insulin Resistance; Bariatric Surgery; Gastric Banding; Gastric Bypass
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Surgery: Obese adult men and women who are undergoing bariatric surgery (gastric bypass or gastric banding).
  Interventions: Procedure: Gastric bypass; Procedure: Gastric banding

INTERVENTIONS:
Procedure: Gastric bypass — NOTE: Surgery will not be paid by the study
  Other Names: GBP
Procedure: Gastric banding — NOTE: Surgery will not be paid by the study
  Other Names: GB

SUMMARY:
This project will study the effects of surgery for obesity on bone metabolism and hormones that regulate appetite.

DETAILED DESCRIPTION:
Subjects will be recruited from the outpatient obesity and surgical clinics at Columbia-Presbyterian Medical Center after they have chosen to undergo a surgical procedure. The groups will not be randomized. Rather, they will decide on their choice of surgery along with their physicians. The patients will be evaluated pre-operatively and followed post-operatively for 5 years.

Initial evaluation will include a complete history and physical examination, measurement of calcium, parathyroid hormone (PTH) and vitamin D, and assessment of skeletal health using markers of bone turnover and bone mineral density.

ELIGIBILITY:
Inclusion criteria:

1. Adult male or female > 18 years of age
2. Scheduled to undergo bariatric surgery

Exclusion criteria:

1. Vitamin D deficiency
2. Primary hyperparathyroidism
3. Treatment with lithium or thiazide diuretics which may alter PTH levels
4. Osteomalacia
5. Untreated hyperthyroidism, liver disease, Cushing's syndrome, rheumatoid arthritis, myeloma or Paget's disease
6. Impaired renal function (serum creatinine >2.0mg/dl) or history of renal osteodystrophy
7. Use of any anti-obesity medications for over 2 weeks 90 days prior to study
8. Participation in any research study 90 days prior to study
9. Any malabsorption syndromes such as celiac sprue
10. Previous bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the outpatient obesity and surgical clinics at Columbia-Presbyterian Medical Center after they have chosen to undergo a surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2003-03-17 (Actual); Primary Completion 2018-11-04 (Actual); Study Completion 2018-11-04 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 5 years
  linear mixed model analysis will be used to study change over time and between surgery

CONTACTS AND LOCATIONS:
Overall Officials: Judith Korner, MD,PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided